CLINICAL TRIAL: NCT01708733
Title: An Evaluation of the Extract of KUAN SIN YIN on Hepatitis C: a Randomized, Double-blinded and Placebo-controlled Clinical Trial.
Brief Title: The Effect of Chinese Herbal Formula (KSY) on HCV Carrier With Abnormal Liver Function
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, Chung-Hua Hsu, chief medical officer, Taipei City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 101001-62-010
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Liver Function
Keywords: HCV carrier; Chinese herbal medicine; Liver function; HCV RNA titer

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- KSY diluted (Placebo Comparator): KSY diluted, 100mg decoction by mouth per day for 6 weeks
- KSY (Experimental): KSY, 100mg decoction by mouth per day for 6 weeks
  Interventions: Drug: KSY

INTERVENTIONS:
Drug: KSY — Chinese herbal formula
  Arms: KSY

SUMMARY:
The aim of the study is to examine whether the Chinese herbal formula (KSY) is effective on HCV Carrier With Abnormal Liver Function.

DETAILED DESCRIPTION:
percentage of change on HCV RNA titer and liver function (GPT).

ELIGIBILITY:
Inclusion Criteria:

* 40 < GPT <200 HCV carrier Age: 18-65 yrs old

Exclusion Criteria:

* Creatinine >2.0 mg/dL Total bilirubin > 2.0mg/dL Not suitable patients diagnosis by physician in charge.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-08; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
HCV RNA titer | 6 weeks

SECONDARY OUTCOMES:
Serum GPT level | 6 weeks

OTHER OUTCOMES:
WHOQOL-BREF | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei City Hospital, Taipei, Taiwan, Taiwan